CLINICAL TRIAL: NCT02354378
Title: A Pilot Study to Assess the Amnesic Properties of Dexmedetomidine in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, Keira Mason, Keira Mason, MD, Boston Children's Hospital
Other Study IDs: IRB-P00004739
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-10

CONDITIONS: Memory; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children undergoing sedation with Dexmedetomidine: Children who will undergo sedation for MRI will be given a memory encoding task during dexmedetomidine bolus induction to measure the effects of sedation. The mere task of naming a picture will encode that picture into memory. When the anesthesia has worn off (at approximately 1 hour later), children will be given a memory recognition task to measure the amnesic effects of dexmedetomidine.
  Interventions: Drug: Dexmedetomidine; Other: Memory Test
- Children not undergoing sedation: A control group of children of similar age scheduled for MRI will be recruited to perform memory recognition testing.
  Interventions: Other: Memory Test

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Precedex
  Groups: Children undergoing sedation with Dexmedetomidine
Other: Memory Test

SUMMARY:
The goal of this study is to determine the effects of dexmedetomidine on memory and recall of children who are receiving dexmedetomidine sedation administered for magnetic resonance imaging (MRI) studies. Dexmedetomidine is currently the standard drug for sedation for diagnostic (MRI, computerized tomography (CT) and Nuclear Medicine) radiological studies at Boston Children's Hospital (BCH). The effect of dexmedetomidine on memory and recall in children has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be between 4 and 14 yrs of age and be undergoing a therapeutic or diagnostic procedure with or without sedation
* The patient must be able to comprehend and perform the task (naming pictures)
* The patient must have a minimum weight of 8 kg

Exclusion Criteria:

* Allergy to Dexmedetomidine (for those patients requiring sedation)
* Procedure of short duration (< 15 min)
* Pregnancy
* Recent use (within 5 half-lives) of centrally acting medications that could affect concentration (e.g. diphenhydramine)

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between the ages of 4 and 14 years old either requiring sedation or attempting without sedation for MRI imaging will be offered inclusion in the study. Sedation will be administered per established and approved BCH sedation guidelines: over 10 minutes, a bolus of 2 mcg/kg of dexmedetomidine will be administered intravenously. The sedation process will not change for this study. During the bolus, pictures will be shown to the child who will be encouraged to name the item in the picture.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2012-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keira Mason, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Mason KP, Kelhoffer ER, Prescilla R, Mehta M, Root JC, Young VJ, Robinson F, Veselis RA. Feasibility of measuring memory response to increasing dexmedetomidine sedation in children. Br J Anaesth. 2017 Feb;118(2):254-263. doi: 10.1093/bja/aew421. PMID 28100530

RESULTS

PARTICIPANT FLOW:
Groups:
- Children Undergoing Sedation With Dexmedetomidine: Children who will undergo sedation for MRI will be given a memory encoding task during dexmedetomidine bolus induction to measure the effects of sedation. The mere task of naming a picture will encode that picture into memory. When the anesthesia has worn off (at approximately 1 hour later), children will be given a memory recognition task to measure the amnesic effects of dexmedetomidine.
  Dexmedetomidine
  Memory Test
- Children Not Undergoing Sedation: A control group of children of similar age scheduled for MRI will be recruited to perform memory recognition testing.
  Memory Test
Period: Overall Study
Arm/Group | Children Undergoing Sedation With Dexmedetomidine | Children Not Undergoing Sedation
Started | 64 | 20
Completed | 30 | 16
Not Completed | 34 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Children Undergoing Sedation With Dexmedetomidine | Children Not Undergoing Sedation | Total
Number analyzed (Participants) | 30 | 16 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 16 | 46
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.1 (1.2) | 9.5 (1.9) | 7.7 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 8 | 30
  Male | 8 | 8 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 16 | 46

OUTCOME MEASURES:

1. Primary Outcome: Sedation Threshold
Description: During the 10-minute bolus infusion of Dexmedetomidine, children will be presented with pictures at 5-second intervals and asked to name the picture. They will be asked to name each picture (e.g., cat, tree, pencil, etc.). A valid response is naming of the picture within 5 seconds, either correctly or incorrectly.The important response measure is whether the child is awake enough to perform the naming task.
Time Frame: Until the child has reviewed cards and is under sedation or for the control group has reviewed 100 cards
Measure: Mean (Standard Deviation); unit: Number of Memory Cards
Arm/Group | Children Undergoing Sedation With Dexmedetomidine | Children Not Undergoing Sedation
Number analyzed (Participants) | 30 | 16
Number of Memory Cards | 26.8 (7.9) | 38.9 (5.9)

2. Secondary Outcome: Memory Threshold
Description: At the presentation of each picture, the child will be asked whether or not he/she remembers having seen it previously. Each response will be coded as correct (true positives and true negatives) or incorrect (false positives and false negatives)
Time Frame: Until 100 cards have been presented to the child. Approx. 10 minutes.
Measure: Mean (Standard Deviation); unit: Number of Memory Cards seen before scan
Arm/Group | Children Undergoing Sedation With Dexmedetomidine | Children Not Undergoing Sedation
Number analyzed (Participants) | 30 | 16
Number of Memory Cards seen before scan | 35.1 (6.6) | 50 (0)

ADVERSE EVENTS:
Arm/Group | Children Undergoing Sedation With Dexmedetomidine | Children Not Undergoing Sedation
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/20
Other Adverse Events (participants affected / at risk) | 0/64 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No